CLINICAL TRIAL: NCT02057952
Title: RCT of Video-Conference & In-Person Weight Loss Services for Adult CHC Patients
Brief Title: HealthyMe Online Weight Management Education/HealthyMe at Home
Acronym: HOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Regenstrief Institute, Inc. (Other); Wishard Health Services (Other)
Responsible Party: Principal Investigator, Daniel Clark, Associate Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1201007860; NIDDK (Other Grant/Funding Number: DK092377)
Record Dates: First submitted 2012-04-06; First posted 2014-02-07 (Estimated); Results first posted 2017-10-27 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Diabetes
Keywords: Weight Management; Diabetes; Exercise; Portion Control; Multiple Chronic Conditions
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity; Multiple Chronic Conditions | interventions — Educational Status; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual Care Control (No Intervention): No intervention.
- In Person Weight Management (Active Comparator): Education and exercise in a community health center environment.
  Interventions: Behavioral: Education and exercise
- Video Conference Weight Management (Experimental): Education and exercise delivered through video conference.
  Interventions: Behavioral: Education and exercise

INTERVENTIONS:
Behavioral: Education and exercise — The active groups will meet twice a week for 75 minutes over six months. They will be followed for an addition six months to monitor maintenance.
  Arms: In Person Weight Management; Video Conference Weight Management

SUMMARY:
The main objective for this project is to identify effective methods of treating obesity in at-risk populations. The investigators will be comparing weight loss from usual care, in person, and video conference weight loss programs. The investigators will follow 210 participants for 12 months to see if they lose and maintain 2kg of weight. The investigators will also compare the costs of video conference versus in person administered programs.

Potentially eligible participants will be identified based on data in the Regenstrief Medical Records System or by referral from the Wishard HealthyMe weight loss program staff or a Wishard Community Health Center (CHC) primary care provider. The PBRN staff will carry-out initial recruitment. Following consent, a baseline assessment will be performed and each participant will be randomized into one of three groups: usual care control, in person weight loss or online video conference weight loss. At 6 and 12 months a follow up assessment will be performed and compared to measures from the investigators baseline assessment. Total costs for each program will be compared as well.

The weight loss interventions involve group meetings two times per week where education, exercise, and social support are provided. Participants will also receive a detailed education booklet. Those randomized to the in-person group will meet in the CHC and those in the video-conference group will meet online in a multi-party video-conference. All participants will receive usual CHC care.

DETAILED DESCRIPTION:
Recruitment will occur in person or by phone by the Practice Based Research Network (PBRN). Prior to recruitment, patients will have been identified as potentially eligible by having a BMI of ≥30<50, age 40-64 years, Community Health Center visit within 12 months and no type 2 diabetes, psychosis or bipolar disorder, current cancer treatment or medication prescriptions for drugs that may unduly influence weight. All of this would be determined from the Regenstrief Medical Records System, by referral from HealthyMe staff, or a CHC primary care provider. Potentially eligible persons must then be approved for the study and moderate-intensity exercise by their primary care provider before the recruitment call and screener from the PBRN. The screener assesses other eligibility criteria such as recent weight loss program enrollment, current physical activity level, residence plans, phone availability, etc. Those who are eligible and initially interested will be referred to the study staff.

Staff will call, describe the study and arrange for an in-home appointment with the potential participant. At the participant's home, the staff will again describe the study and consent the participant. The first assessment will take place at this time. The baseline assessment pertains of demographic questions, living situation questions, smoking status, weight history, Patient Health Questionnaire (PHQ), New Vital Sign (NVS) Nutrition Literacy and Numeracy Survey, the Subjective Numeracy Scale, Short Form 36, Social Support and Exercise, Social Support and Eating Habits, Exercise enjoyment scales, Wellness Evaluation of Lifestyle (WEL), low fat diet efficacy scale, exercise self efficacy scale, and an online dietary recall (ASA 24) provided by the National Cancer Institute as well as blood pressure, weight, height and waist circumference. They will also be asked to wear an armband accelerometer for two weeks to let the staff know how much energy they are expending.

The participants will be randomized to three different arms: usual care, in center education and exercise, or education and exercise via video conference. The attached handouts, placemats, as well as portion control dinnerware will be given to the active arms of the study. The sessions for both groups will occur twice a week for approximately 75 minutes. Those randomized to the video conference arm will have a computer with Internet access installed in their home. All Internet related expenses will be covered by the study during the duration of the classes and the computer will be removed at the end of the study.

Sessions for the two active arms will occur twice per month in months 6-9 and once a month for months 10-12. They will include an exercise and educational portion to last about 75 minutes.

We will be measuring change in weight, body measurements and improvements in the NVS at six months and have a final assessment at 12 months. They will again be asked to wear the accelerometer for two weeks and to answer the questions in the attached survey. Their weight and blood pressure will again be recorded.

During the course of the study, participants may need to be called to set up appointments, remind them of sessions or assist them with their equipment.

ELIGIBILITY:
Inclusion Criteria:

* One or more community health visits in the past 12 months
* Body mass index (BMI) of ≥30<50
* English Speaking
* Access to a telephone
* A residence
* Willingness to be randomized
* Willingness to have a computer installed in the home
* Weight loss referral from CHC provider

Exclusion Criteria:

* Current diagnosis of type 2 diabetes
* Current treatment for cancer
* Current diagnosis of psychosis or bipolar disorder
* Illness that might be associated with weight change, such as asthma, (because of treatment with corticosteroids), psychosis
* Use of medications that might cause weight gain or loss such as hypoglycemic oral medicines or insulin, corticosteroids, some anti-depressants, weight loss medications
* Unwilling or unable to provide informed consent
* Receiving disability insurance
* Pregnant or nursing in the past six months, or plans to become so within 12 months
* Residence outside of Marion County, Indiana
* Residence relocation plans within 12 months
* Enrolled in weight loss program within past 6 months
* Meeting physical activity guidelines
* Planned or prior bariatric surgery
* Substance abuse
* History of treatment for eating disorder
* Unstable weight gain or loss of ≥5% in the last 3 months

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2012-04; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel O. Clark, Ph.D, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Shell AL, Hsueh L, Vrany EA, Clark DO, Keith NR, Xu H, Stewart JC. Depressive symptom severity as a predictor of attendance in the HOME behavioral weight loss trial. J Psychosom Res. 2020 Apr;131:109970. doi: 10.1016/j.jpsychores.2020.109970. Epub 2020 Feb 15. PMID 32088427

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care Control | In Person Weight Management | Video Conference Weight Management
Started | 51 | 49 | 50
Completed | 43 | 39 | 28
Not Completed | 8 | 10 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care Control | In Person Weight Management | Video Conference Weight Management | Total
Number analyzed (Participants) | 51 | 49 | 50 | 150
Age, Continuous [Mean (Standard Deviation); unit: YEAR OF AGE] | 53.9 (6.1) | 53.2 (8.1) | 53.2 (6.1) | 53.4 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 38 | 46 | 123
  Male | 12 | 11 | 4 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 2
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 49 | 49 | 50 | 148
Region of Enrollment [Number; unit: participants]
  United States | 51 | 49 | 50 | 150
Years of Education, continuous [Mean (Standard Deviation); unit: Years] | 13.2 (2.4) | 13.6 (2.4) | 12.6 (1.7) | 13.1 (2.2)
weight, continuous [Mean (Standard Deviation); unit: pounds] | 236.4 (43.6) | 234.1 (46.7) | 227.6 (35.5) | 232.7 (42.0)
body mass index, continuous [Mean (Standard Deviation); unit: kilograms divided by meters squared] | 39.4 (6.2) | 38.9 (5.8) | 38.5 (5.5) | 38.9 (5.8)
Short Form 36 (RANGE 0 [Worst] -100 [Best]), continuous [Mean (Standard Deviation); unit: standardized score] | 52.8 (19.0) | 59.2 (18.4) | 56.5 (21.8) | 56.1 (19.8)
Patient Health Questionnaire (range 0 [best] -27[worst]), continuous [Mean (Standard Deviation); unit: standardized score] | 7.6 (6.0) | 6.9 (5.5) | 7.3 (5.3) | 7.3 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: Body Weight
Description: Change in weight from baseline to 12 months reported in pounds.
Time Frame: Baseline to 12 Months
Population: The number of participants analyzed is based on the number of participants who completed weight data at baseline and 12 months.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Usual Care Control | In Person Weight Management | Video Conference Weight Management
Number analyzed (Participants) | 43 | 39 | 28
pounds | -0.8 (10.9) | -1.5 (14.6) | -7.3 (11.5)

2. Primary Outcome: Attendance Reported in Minutes
Description: Minutes of participation in study sessions.
Time Frame: 12 Months
Population: Usual care participants didn't have access to the experimental treatments. In person and video conference arm participants were all eligible for participation.
Measure: Median (Full Range); unit: minutes
Arm/Group | Usual Care Control | In Person Weight Management | Video Conference Weight Management
Number analyzed (Participants) | 0 | 49 | 50
minutes |  | 0 [0 to 2880] | 90 [0 to 2640]

3. Primary Outcome: Change in Body Weight From Baseline to 6 Months.
Description: Change in body weight from baseline to 6 months.
Time Frame: 12 months
Population: Analysis are based on number of participants with complete weight data at baseline and 6 months.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Usual Care Control | In Person Weight Management | Video Conference Weight Management
Number analyzed (Participants) | 49 | 42 | 33
pounds | 1.3 (9.8) | -0.9 (10.7) | 3.1 (9.2)

4. Secondary Outcome: Change in Short Form 36 Survey Score
Description: The Short Form 36 survey or Short-Form 36 is a patient report survey. Scores range from 0 (worst) to 100 (best) and represent overall health-related quality of life.
Time Frame: Baseline to 12 Months
Population: The analysis of change based on participants with complete Short Form 36 (SF36) scores at baseline and 12 months.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Usual Care Control | In Person Weight Management | Video Conference Weight Management
Number analyzed (Participants) | 43 | 39 | 28
score on scale | 6.5 (8.7) | -3.1 (18.3) | 7.1 (19.6)

5. Secondary Outcome: Change in Systolic Blood Pressure
Description: Systolic blood pressure. Measured using blood pressure cuff and sphygmomanometer. Units in Milometers of Mercury (mmHg). Scale range is based on participants' actual blood pressure (change baseline to 12 months). Negative value indicates decrease in blood pressure.
Time Frame: 12 Months
Population: Participants who completed 12 month follow-up
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Usual Care Control | In Person Weight Management | Video Conference Weight Management
Number analyzed (Participants) | 40 | 36 | 26
mmHg | -3.8 (14.6) | -1.1 (17.2) | -7.4 (19.8)

6. Secondary Outcome: Cost-effectiveness
Description: The cost effectiveness ratios were calculated by dividing the difference in total cost per arm by the difference in percent of subjects with 2+ kg weight loss
Time Frame: 12 months
Measure: Number; unit: Total Cost / 100 participants
Arm/Group | Usual Care Control | In Person Weight Management | Video Conference Weight Management
Number analyzed (Participants) | 51 | 49 | 50
Total Cost / 100 participants | 0 | 5564 | 3744

7. Secondary Outcome: Change in SF 36 From Baseline to 6 Months
Description: as for outcome 4
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care Control | In Person Weight Management | Video Conference Weight Management
Number analyzed (Participants) | 49 | 42 | 32
units on a scale | 3.5 (15.6) | -1.1 (13.5) | 6.1 (13.6)

8. Secondary Outcome: Change in Systolic Blood Pressure
Description: Change in pressure from baseline to 6 months
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Usual Care Control | In Person Weight Management | Video Conference Weight Management
Number analyzed (Participants) | 43 | 38 | 32
mmHg | 2.5 (15.1) | -0.8 (18.9) | 7.4 (20.5)

9. Secondary Outcome: Change in Diastolic Blood Pressure at 6 Months
Description: Change in pressure from baseline to 6 months
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Usual Care Control | In Person Weight Management | Video Conference Weight Management
Number analyzed (Participants) | 43 | 38 | 32
mmHg | 1.8 (10.4) | 0 (12.5) | 6.0 (19.7)

10. Secondary Outcome: Change in Diastolic Blood Pressure Baseline to 12 Months
Description: Diastolic blood pressure change from baseline to 12 months. Measured using blood pressure cuff and sphygmomanometer. Units in Milometers of Mercury (mmHg). Scale range is based on participants' actual blood pressure (change baseline to 12 months; negative value indicates decrease in blood pressure).
Time Frame: 12 Months
Population: Participants who completed 12 month follow-up
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Usual Care Control | In Person Weight Management | Video Conference Weight Management
Number analyzed (Participants) | 40 | 36 | 26
mmHg | -5.8 (11.4) | -2.6 (11.8) | -8.1 (20.2)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Usual Care Control | In Person Weight Management | Video Conference Weight Management
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/49 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/49 | 0/50
Other Adverse Events (participants affected / at risk) | 0/51 | 0/49 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2015-08-13): https://cdn.clinicaltrials.gov/large-docs/52/NCT02057952/Prot_000.pdf
  • Statistical Analysis Plan (2015-08-13): https://cdn.clinicaltrials.gov/large-docs/52/NCT02057952/SAP_001.pdf
  • Informed Consent Form (2015-08-24): https://cdn.clinicaltrials.gov/large-docs/52/NCT02057952/ICF_002.pdf